CLINICAL TRIAL: NCT02079493
Title: Prospective Functional Outcome Study of the Knee
Acronym: PFOSK
Status: Terminated | Type: Observational
Why Stopped: Not enough subject enrollment
Sponsor: Tufts Medical Center (Other)
Collaborators: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 11109-Conformis
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee replacement; functional testing
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Knee Arthroplasty patients: TKA patients
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Knee replacement
  Other Names: ConforMIS, Off the shelf, TKA

SUMMARY:
The purpose of this study is to obtain patient-oriented and clinically-oriented physical function outcomes both pre-operatively and post-operatively in patients receiving a total knee arthroplasty .

DETAILED DESCRIPTION:
This study aims to use up to 75 patients at 3 centers to determine a baseline short-term postoperative physical function status of patients undergoing a total knee arthroplasty through patient and clinically based assessments. The KOOS score will collect data on the patient's physical function, stiffness, and pain. The BERG balance, TUG, and TUDS tests will be used quantitatively to assess the patient's ability to conduct activities of daily living like walking for an extended period of time, standing from a seated position, and maintaining balance while performing a series of actions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or non-pregnant female age 18 years or older at time of study
* Patient is a candidate for a total knee arthroplasty
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with a primary diagnosis other than osteoarthritis of the knee as determined by an orthopaedic surgeon
* Patients who have had any previous lower extremity procedure
* Patients with a BMI greater than or equal to 40
* Patients with an active infection within the affected knee joint Patients with a neuromuscular or neurosensory deficiency that may limit the ability of the patient to evaluate the safety and efficacy of the device
* Patient is diagnosed with systemic disease or metabolic disorder leading to progressive bone deterioration (e.g. Lupus Erythematosus, Paget's Disease)
* Patient is immunologically suppressed or receiving chronic steroids in excess of normal physiological requirements (e.g. greater than 30 days)
* Patient has a known sensitivity to device materials
* Non-English speaking patients
* Patient is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total knee arthroplasty patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Functional testing | 6 weeks post-op
  Assess patient functional outcomes
Functional testing | 6 months post-op
  Assess patient functional outcomes
Functional testing | 1-year post-op
  Assess patient functional outcomes

SECONDARY OUTCOMES:
Outcome questionnaires | 6-weeks post-op
  to assess knee pain and function
Outcome questionnaires | 6-months post-op
  to assess knee pain and function
outcome questionnaires | 1-year post-op
  to assess knee pain and function

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Smith, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Due to PI moving locations and site closing out study, not all follow-up data will be collected and results will not be analyzed